CLINICAL TRIAL: NCT04334005
Title: Effect of Vitamin D Administration on Prevention and Treatment of Mild Forms of Suspected Covid-19
Brief Title: Vitamin D on Prevention and Treatment of COVID-19
Acronym: COVITD-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Manuel Castillo Garzón, MD, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVITD-19
Record Dates: First submitted 2020-03-29; First posted 2020-04-03 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Patients Infected With COVID-19
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Prescription of NSAIDs, ACE2 inhibitor, ARB or thiazolidinediones, according to clinician criteria, based on the current recommendations.
  Interventions: Dietary Supplement: Vitamin D
- Intervention group (Experimental): 25000 UI of vitamin D supplement in addition to the above-mentioned drug recommendations.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — The intervention group will receive a single dose of 25000 UI of vitamin D supplement in addition to prescription of NSAIDs, ACE2 inhibitor, ARB or thiazolidinediones, according to clinician criteria, based on the current recommendations. Vitamin D supplementation will be taken in the morning together with a toast with olive oil to facilitate its absorption.

SUMMARY:
The new outbreak of the SARS-CoV-2 coronavirus is causing an important pandemic affecting a large number of people all-over the world. Vitamin D is a hormone precursor produced by our own body with the help of sunlight which has an important role on adaptive immunity and cellular differentiation, maturation and proliferation of several immune cells. Reduced levels of vitamin D in calves were positioned as the main cause of bovine coronavirus infection in the past. Therefore, it seems plausible that the use of vitamin D as a nutritional ergogenic aid could be a potential intervention to fight against COVID-19 infected patients which remain asymptomatic or which have non-severe and severe symptoms. This study aims to investigate whether the use of vitamin D as an immune modulator agent induces significant improvements of health status and outcomes in non-severe symptomatic patients infected with COVID-19 as well as preventing COVID-19 health deterioration. We hypothesize that vitamin D will significantly improve hard endpoints related to COVID-19 deleterious consequences compared with a usual care control group.

ELIGIBILITY:
Inclusion Criteria:

* Non-severe symptomatic patients who present cough, fever, nasal congestion, gastrointestinal symptoms, fatigue, anosmia, ageusia or alternative signs of respiratory infections.

Exclusion Criteria:

* Patients presenting severe respiratory and/or multisystemic symptoms compatible with advanced COVID-19 and intercurrent acute or severe chronic diseases (i.e. active cancer).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-10 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite of cumulative death (i.e. mortality) for all causes and for specific causes. | Through study completion, an average of 10 weeks

SECONDARY OUTCOMES:
Necessity of invasive assisted ventilation | Through study completion, an average of 10 weeks
Necessity of non-invasive assisted ventilation | Through study completion, an average of 10 weeks
Intensive care unit admission | Through study completion, an average of 10 weeks
Post-anesthesia care unit admission | Through study completion, an average of 10 weeks
Hospital admission | Through study completion, an average of 10 weeks
Medical consultation | Through study completion, an average of 10 weeks
Home care and isolation time | Through study completion, an average of 10 weeks
Bed rest time | Through study completion, an average of 10 weeks
symptoms' duration (i.e. cough, fever, nasal congestion, gastrointestinal symptoms, fatigue, anosmia, ageusia, diarrhea or alternative signs of COVID-19) | Through study completion, an average of 10 weeks
Subjective perception of recovery | Through study completion, an average of 10 weeks
  It will be measure by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Manuel J Castillo, MD, PhD, Principal Investigator — Universidad de Granada
Locations (2):
- Spain (2):
  - Universidad de Granada, Granada, Andalusia
  - Medicine Faculty, Granada

IPD SHARING:
Plan to Share IPD: Undecided